CLINICAL TRIAL: NCT06909045
Title: Randomized Controlled Trial Comparing Adaptive Versus Continuous Subthalamic Nucleus Deep Brain Stimulation in Parkinson's Disease
Brief Title: Adaptive vs. Continuous Subthalamic Nucleus Deep Brain Stimulation in Parkinson's Disease
Acronym: CLOSE-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: HagaZiekenhuis (Other); Maastricht University Medical Center (Other); Universitair Ziekenhuis Leuven (Unknown)
Responsible Party: Principal Investigator, dr. Martijn Beudel, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL009220
Record Dates: First submitted 2025-03-10; First posted 2025-04-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Deep Brain Stimulation; Parkinson Disease
Keywords: adaptive DBS; continue DBS; aDBS; cDBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aDBS group (Experimental): 65 patients with Parkinson's disease will receive adaptive DBS.
  Interventions: Other: Adaptive DBS
- cDBS group (Active Comparator): 65 patients with Parkinson's disease will receive continue DBS.
  Interventions: Other: Continue DBS

INTERVENTIONS:
Other: Adaptive DBS — The Medtronic Percept device will be activated with the aDBS functionality. Participant will receive adaptive DBS.
  Arms: aDBS group
Other: Continue DBS — The Medtronic Percept device will be equipped with aDBS functionality (to maintain the blinding of the allocation), but this functionality will remain inactive. Participant will receive continue DBS.
  Arms: cDBS group

SUMMARY:
The objective of the CLOSE-PD study is to compare the efficacy of adaptive deep brain stimulation (aDBS) with continue deep brain stimulation (cDBS) in patients with Parkinson's disease. The main question it aims to answer is:

- whether the change in daily mean ON time without troublesome dyskinesia in aDBS is greater than cDBS over a six-month follow-up period?

Researchers will compare aDBS to regular continue deep brain stimulation (cDBS).

Participants will:

* be set up to cDBS during the first programming visit (visit 2);
* be randomized 1:1 to aDBS or cDBS two weeks after visit 2;
* follow-up will be at three and six months after visit 2;
* complete PD Home diary at baseline, two weeks, three months and at six months after visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD based on the UK Brain Bank criteria (Hughes et al. 1992);
* Age older than 18 years;
* Previous implantation of Medtronic PerceptTM PC/RC DBS electrodes bilateral targeting the STN;
* Optimal contact point compatible with aDBS in at least one STN;
* Reliable beta peak in at least one STN;
* Able to provide informed consent and comply with the study protocol;
* Understand the Dutch language.

Exclusion Criteria:

* Legally incompetent adults;
* Patients with ongoing participation in other clinical trials involving neurological interventions;
* Inability to recognize the difference between the motor ON or OFF state;
* Mild cognitive impairment or dementia;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Home PD diary | change from baseline to six months of DBS
  The primary outcome is the comparison between the aDBS group and the cDBS group of the change from baseline to six months in mean daily ON time without troublesome dyskinesia. Daily ON time without troublesome dyskinesia is measured with the PD home diary. The PD home diary is a self-reported tool for tracking motor symptoms in Parkinson's patients every 30 minutes for three days within a one-week window

SECONDARY OUTCOMES:
PD Home diary | during six months of follow-up
  ON time without troublesome dyskinesia
PD Home diary | during six months of follow-up
  ON time with troublesome dyskinesia
PD Home diary | during six months of follow-up
  ON time without dyskinesia
PD Home diary | during six months of follow-up
  OFF time
PD Home diary | during six months of follow-up
  Asleep time
MDS-UPDRS III (ON and OFF phase) | change from baseline to six months of DBS
  Motor symptoms
MDS-UPDRS IV | change from baseline to six months of DBS
  Motor complication including motor fluctuations and dyskinesias
Academic Medical Center Linear Disability Score (ALDS) (ON and OFF phase) | change from baseline to six months of DBS
  Level of physical disability
Parkinson's Disease Questionnaire 39 (PDQ-39) | change from baseline to six months of DBS
  Quality of life
Dopaminergic medication usage | during six months of follow-up
Montreal Cognitive Assessment (MoCA) | change from baseline to six months of DBS
  MoCA is a cognitive screening tool for detecting and scoring cognitive impairment
Beck Depression Inventory (BDI) | change from baseline to six months of DBS
  Mood status
Starkstein Apathy Scale (SAS) | change from baseline to six months of DBS
  Apathy status
Parkinson's Disease Sleep Scale (PDSS-2) | during six months of follow-up
  Sleep disturbances and quality of sleep
Side effects | during six months of follow-up
  Number and sort of side effects
Time of DBS titration | during six months of follow-up
  Duration of DBS titration based on the number and duration of hospital visits
Time to final adjustment of the DBS settings | during six months of follow-up
  first time point for stimulation parameters following the last adjustment of the stimulation parameters
Assessor's evaluation of the ease of programming | after six months of follow-up
  Five-point Likert scale
Beta oscillatory activity | during six months of follow-up
  Amount of decrease of oscillatory activity in the beta range
DBS settings (1) | during six months of follow-up
  Electrical energy consumption expressed by the Total electrical energy delivered (TEED)
DBS settings (2) | during six months of follow-up
  DBS amplitudes in mA
DBS settings (3) | during six months of follow-up
  Average stimulation fraction expressed as percentages
LFP characteristics (2) | during six months of follow-up
  Beta power spectral density expressed as µV²/Hz
LFP characteristics (2) | during six months of follow-up
  Beta volatility expressed as a.u.
Participant's evaluation of the burden of the treatment | after six months of follow-up
  Five-point Likert scale
Participant's satisfaction on the outcome of treatment | after six months of follow-up
  Five-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Beudel, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (4):
- UZ Leuven, Leuven, Belgium
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Maastricht UMC+, Maastricht
  - HagaZiekenhuis, The Hague

IPD SHARING:
Plan to Share IPD: Yes
Upon request, IPD will be shared through restricted access via a secure online database.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It will be available two years after the results are published.